CLINICAL TRIAL: NCT03668847
Title: A Phase II: Safety and Tolerance of 4-Demethyl-4-cholesteryloxycarbonylpenclomedine (DM-CHOC-PEN) in Adolescent and Young Adults (AYA) With Malignancies Involving the CNS
Brief Title: DM-CHOC-PEN for Brain Tumors in AYA Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DEKK-TEC, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTI-026
Record Dates: First submitted 2018-09-05; First posted 2018-09-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Advanced Cancer; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DM-CHOC-PEN (Experimental): 4-Demethyl-4-cholesteryloxycarbonylpenclomedine (DM-CHOC-PEN) - 75 or 98.7 mg/m2 emulsion will be administered IV once every 21-days until relapse
  Interventions: Drug: DM-CHOC-PEN

INTERVENTIONS:
Drug: DM-CHOC-PEN — DM-CHOC-PEN administration by IV infusion

SUMMARY:
4-Demethyl-4-cholesteryloxycarbonylpenclomedine (DM-CHOC-PEN) is a polychlorinated pyridyl cholesterol carbonate that is lipophilic, electrically neural, crosses the blood brain barrier (BBB), ability to localize in intracranial tumor tissue, lacks neurotoxicity and not transported out of the brain via Pgp (p-glycoprotein). DM-CHOC-PEN has completed a Phase I Adolescent and Young Adult (AYA) trial in humans, some of which possessed primary and secondary tumors involving the brain. Complete remissions in both primary (astrocytoma, GBM) and metastatic lung cancers were reported.

This Phase II trial is closed for adolescent and young adults (AYA) subjects with advanced cancer - brain involvement is required.

DETAILED DESCRIPTION:
The primary goal of this Phase II AYA oncology clinical trial was to evaluate the safety and efficacy of 4-demethyl-4-cholesteryloxycarbonylpenclomedine (DM-CHOC-PEN), as anticancer therapy in AYA individuals with advanced cancer involving the central or spinal nervous system (CNS & SNS).

DM-CHOC-PEN is a polychlorinated pyridine cholesteryloxycarbonate that crosses the blood brain barrier (BBB), accumulates in CNS tumor tissue in humans and has produced objective responses, with acceptable/reversible hepatic toxicities (in patients with prior liver disease) and no evidence of hematological, renal, neuro-toxicities with improved quality of life and overall survival in adolescent, young adult and adult Phase I/II clinical trials - IND - 68,876.

The FDA has supported the Phase II clinical trial designed to identify safety and efficacy in AYA cancers subjects and the trial has been completed with acceptable toxicity and MTDs identified.

Almost 700,000 people in the US are living with tumors involving the CNS or spinal nervous system (SNS) tumors. Nearly 15% of these tumors involve the adolescent/young adult (AYA) population, aged 15-39 years of age. It is predicted that 10,617 AYA individuals will be diagnosed with brain or CNS tumors resulting in 434 deaths this year in the US. Trends in CNS tumors have sharply increased since 1989 for AYA individuals with a history of cancer, who appeared to have 'beaten the odds', only to have a re-occurrence from cancer involving the CNS after years of remission; the most common types of cancer in AYA individuals are - melanoma, leukemia and sarcomas. This group of individuals deserves special attention.

For males and female individuals <20 years of age, primary brain and secondary cancers of the CNS and spinal nervous system (SNS) are the most common causes of death from cancer and in the 20-39 year age group the first cause of cancer-related deaths in males and the fifth cause of cancer-related deaths in females. The incidence and histology of cancer types does vary according to subject age.

A critical component in designing an agent that will cross the protective blood brain barrier (BBB) is that the agent must be readily transported intracerebrally, does not produce local irritation/neurotoxicity and is not recycled back into the general circulation. After IV administration DM-CHOC-PEN readily penetrates the BBB, is not a substrate for the transporter protein P-glycoprotein (P-gp) and has shown anticancer activity in CNS tumors. The effective transport of DM-CHOC-PEN into CNS tumors in adults without neurotic behavioral alterations and associated events supports the drug's use in children with CNS tumors at an age in which brain development and maturation is still very active with cognitive lability. The observed responses noted in adults with metastatic cancers involving the CNS and cerebellum treated with DM-CHOC-PEN may also occur in medulloblastoma in AYA. Thus, the drug's unique properties and lack of toxicities noted in the adult studies merits the Phase I trial proposed here in children.

The specific objectives of this Phase I study were to:

1. Conduct a Phase II clinical trial with DM-CHOC-PEN in AYA individuals that have advanced cancers with central or spinal nervous systems involvements and monitor safety and document anticancer activity for the drug. All data was between investigators communicated through an e-RAP program. This was accomplished through IND - 68.876.
2. Verify the pharmacokinetic/dynamic profiles of DM-CHOC-PEN and metabolites in AYA subjects with advanced cancers involving the central nervous system.
3. Analyze data and prepare an Orphan Drug Designated package for FDA submission for AYA subjects with CNS involvement from cancer for review.

ELIGIBILITY:
Inclusion Criteria: was as follows -

* Subjects must have histological proof of a malignancy, which has been treated with standard treatments, which may include radiation, and measurable lesions are not required but must have evidence that the disease is advanced.
* Subjects must have life expectancy of at least 12 weeks and a Karnofsky performance score: > 60 % (or a Zubrod performance status of < 2).
* The age limit - a limit of 39 years of age. Gender is not a criterion.
* All subjects must be off previous chemo- and/or radiotherapy for at least three (3) weeks prior to entrance into the study and have recovered from any toxic effects induced by such treatment(s); no nitrosourea type drug or ipilumimab treatments are permitted within the last six (6) weeks prior to enrollment. No major surgery within 14 days of enrollment. Subjects may continue to receive anti- estrogen/steroid therapy that has been initiated at least eight weeks prior to enrollment in the study.
* Subjects should have adequate bone marrow function defined as a peripheral WBC >3,000/mm3 with an ANC >1500/mm3 and a platelet count >100,000/mm3.
* Subjects should have hepatic function (alkaline phosphatase, AST and ALT) < ULN and renal functions with serum creatinine - <1.5 x UNL. If a patient has liver metastasis and/or a history of liver disease - they will receive a lower dose of the drug per treatment protocol.
* Subjects should not be allergic to eggs or soy beans.
* Subjects must be medically, psychologically and neurologically stable and have triplicate baseline ECG's with a mean QTc interval <500 ms and >300 ms and neither a history of congenital prolonged or short QT syndrome. Subjects with a history of cardiac disease must be stable.
* Subjects and/or legal guardian must understand the nature of the study and be willing to sign an informed consent that complies with the investigator/DEKK-TEC policies and approved by the Human Investigation Review Committee.

Exclusion Criteria: will be as follows:

* Subjects with concurrent severe and/or uncontrolled medical co-morbidities - including active infections, unstable uncontrolled diabetes, cardiovascular and pulmonary, renal, psychiatric or social conditions that could compromise the safety or compliance of treatment are not eligible.
* Concomitant chemotherapy or radiotherapy was not permitted.
* Pregnant or lactating females were excluded. Women of childbearing age, and their sexual partners, must use an effective contraception program. Males who are having sexual relations with women capable of child bearing must use the barrier birth control while on the study and for 3-months after the last dose of the study drug.
* Subjects taking CYP3A4 inducers or inhibitors were not eligible since it is not known whether the study drug is metabolized through this pathway. The following CYP3A4 inhibitors/inducers are not permitted during the trial - phenobarbital, fluconazole, erythromycin, verapamil; the latter 3-drugs are moderate CYP3A4 inhibitors.
* Subjects taking the following medications may experience QT/QTc interval prolongation and are not eligible for the trial - most anti-arrhythmia drugs (incl. amiodarone), erythromycin, quinolone antibiotics, ketoconazole, Zithromax, and phenothiazine and were denied enrollment in the study. The possible interactions of these drugs and DM-CHOC-PEN have not been established.
* Coagulopathies - patients requiring full dose anticoagulation with warfarin were excluded.

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Brain Tumor Responses to Therapy | From date of entry into the study until the date of first documented progression or date of of death from any cause, which ever came first, assessed up to 100 months.
  MRI of the brain

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax], Area Under the Curve [AUC] | From initiation of treatment until end of therapy or death from any cause or which ever comes first, assessed up to 8-months.
  Blood levels for DM-CHOC-PEN and metabolites will be measured before and after each treatment; HPLC procedures will be involved.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Baghian, MD, Principal Investigator — Tulane University Medical Center; Tallat Mahmmod, MD, Principal Investigator — Detroit Clinical Research Center; Marcus L Ware, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Tulane University Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All data regarding subject enrollment will be coded and electronically submitted to DEKK-TEC for submission to the FDA. Other trial sites are being evaluated. After all are chosen a decision will be made.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data summary is being prepared as a manuscript for distribution.
  December 31, 2022
Access Criteria: The requesting individuals must be established investigators.